CLINICAL TRIAL: NCT02847962
Title: Newly Formulated, Extruded Fortified-blended Foods for Food Aid: the MFFAPP Tanzania Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: Project Concern International - Tanzania (Unknown); National Institute for Medical Research, Tanzania (Other Government); United States Department of Agriculture Foreign Agricultural Service (Other)
Responsible Party: Principal Investigator, Brian Lindshield, Associate Professor, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFE-621-2012/033-00
Record Dates: First submitted 2016-07-20; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Anemia, Iron-Deficiency; Deficiency, Vitamin A
Keywords: Fortified-blended foods; Extrusion; Sorghum; Cowpea; Vitamin A; Iron; Protein; Food Aid; Anemia, Iron-Deficiency; Deficiency, Vitamin A; Growth Velocity; Stunting; Wasting; Protein-Energy Malnutrition; Complementary Feeding; Corn; Soy; Fortified Foods; Food assistance
MeSH Terms: conditions — Anemia, Iron-Deficiency; Vitamin A Deficiency; Growth Disorders; Cachexia; Protein-Energy Malnutrition; Callosities | interventions — Placental Lactogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Control (No FBF) (No Intervention): FBF provided after the intervention period
- Corn Soy Blend Plus (CSB+) (Active Comparator): Consumed Corn Soy Blend Plus (CSB+)
  Interventions: Other: Corn Soy Blend Plus (CSB+)
- Corn Soy Blend 14 (CSB14) (Experimental): Consumed Corn Soy Blend 14 (CSB14)
  Interventions: Other: Corn Soy Blend 14 (CSB14)
- White Sorghum Cowpea Blend Variety 1 (Experimental): Consumed White Sorghum Cowpea Blend Variety 1
  Interventions: Other: White Sorghum Cowpea Blend Variety 1
- White Sorghum Cowpea Blend Variety 2 (Experimental): Consumed White Sorghum Cowpea Blend Variety 2
  Interventions: Other: White Sorghum Cowpea Blend Variety 2
- Red Sorghum Cowpea Blend (Experimental): Consumed Red Sorghum Cowpea Blend
  Interventions: Other: Red Sorghum Cowpea Blend
- White Sorghum Soy Blend (Experimental): Consumed White Sorghum Soy Blend
  Interventions: Other: White Sorghum Soy Blend

INTERVENTIONS:
Other: Corn Soy Blend Plus (CSB+)
  Arms: Corn Soy Blend Plus (CSB+)
Other: Corn Soy Blend 14 (CSB14)
  Arms: Corn Soy Blend 14 (CSB14)
Other: White Sorghum Cowpea Blend Variety 1
  Arms: White Sorghum Cowpea Blend Variety 1
Other: White Sorghum Cowpea Blend Variety 2
  Arms: White Sorghum Cowpea Blend Variety 2
Other: Red Sorghum Cowpea Blend
  Arms: Red Sorghum Cowpea Blend
Other: White Sorghum Soy Blend
  Arms: White Sorghum Soy Blend

SUMMARY:
Corn-soy vitamin and mineral fortified blended foods (FBFs) are primarily used for food aid, although sorghum and cowpea may be suitable alternative FBF commodities. The objective of the Micronutrient Fortified Food Aid Pilot Project (MFFAPP) Tanzania Efficacy Study is to determine whether newly formulated, extruded sorghum- and cowpea-based FBFs have equal, or better, nutritive value and acceptance compared to a traditional corn-soy blend. The effectiveness of each blend will be determined in an efficacy study of Tanzanian children under the age of 5 that are deficient, or at risk for deficiency, in iron and vitamin A.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin <10.3mg/dl
* Weight-for-height z-scores >-3

Exclusion Criteria:

* Exclusive breastfeeding
* Unwillingness to travel to health facilities
* Enrollment of child in school during study period
* Anticipated relocation of the family during the study
* Allergy to the fortified-blended food product ingredients

Ages: 6 Months to 53 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2179 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin Change | 0, 10, 20 weeks (baseline, midline, and end line)
Dried blood spot retinol binding protein change | 0, 10, 20 weeks (baseline, midline, and end line)
  Assessment of vitamin A status

SECONDARY OUTCOMES:
Height-for-age change | 0, 10, 20 weeks (baseline, midline, and end line)
Weight-for-age change | 0, 10, 20 weeks (baseline, midline, and end line)
Weight-for-height change | 0, 10, 20 weeks (baseline, midline, and end line)
Moderate malnutrition status change | 0, 10, 20 weeks (baseline, midline, and end line)
  Weight-for-age between -3 and -2 z-scores below the median of the WHO child growth standards
Mid-upper arm circumference change | 0, 10, 20 weeks (baseline, midline, and end line)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delimont NM, Vahl CI, Kayanda R, Msuya W, Mulford M, Alberghine P, Praygod G, Mngara J, Alavi S, Lindshield BL. Complementary Feeding of Sorghum-Based and Corn-Based Fortified Blended Foods Results in Similar Iron, Vitamin A, and Anthropometric Outcomes in the MFFAPP Tanzania Efficacy Study. Curr Dev Nutr. 2019 Apr 10;3(6):nzz027. doi: 10.1093/cdn/nzz027. eCollection 2019 Jun. PMID 31143849
- [Derived] Delimont NM, Chanadang S, Joseph MV, Rockler BE, Guo Q, Regier GK, Mulford MR, Kayanda R, Range M, Mziray Z, Jonas A, Mugyabuso J, Msuya W, Lilja NK, Procter SB, Chambers E 4th, Alavi S, Lindshield BL. The MFFAPP Tanzania Efficacy Study Protocol: Newly Formulated, Extruded, Fortified Blended Foods for Food Aid. Curr Dev Nutr. 2017 Apr 25;1(5):e000315. doi: 10.3945/cdn.116.000315. eCollection 2017 May. PMID 29955700